CLINICAL TRIAL: NCT06919640
Title: Psilocybin With Intracranial Neural Sensing
Acronym: PINS
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Joshua Woolley, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Joshua Woolley, MD, PhD, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-39870; 175145 (Other: FDA); PR#202507H (Other: Research Panel of California)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain
Keywords: chronic pain; psilocybin; psychedelic; pain; dbs
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 10mg oral psilocybin (Experimental)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 10mg oral psilocybin

SUMMARY:
This is an open-label, single-arm, pilot study exploring the neural, sensory, and cognitive effects of a single, medium dose of psilocybin in patients with chronic pain who already have implanted sensing-capable deep brain stimulation (DBS) devices. Outcomes include multi-site neural recording from previously placed ambulatory sensing-capable DBS devices, quantitative sensory and cognitive testing, and self-reports of pain. We hypothesize that psilocybin will change functional connectivity, decrease clinical and task-based pain reports, and improve cognitive functions.

DETAILED DESCRIPTION:
This is an open-label, single-arm, pilot study exploring the neural, sensory, and cognitive effects of a single, medium dose of psilocybin in patients with chronic pain who already have implanted sensing-capable deep brain stimulation (DBS) devices. Outcomes include multi-site neural recording from previously placed ambulatory sensing-capable DBS devices, quantitative sensory and cognitive testing, and self-reports of pain. We hypothesize that psilocybin will change functional connectivity, decrease clinical and task-based pain reports, and improve cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Currently implanted chronic brain sensing device (such as RC+S or Percept)
* Not currently enrolled in another trial
* Ability to speak and read English
* Able to attend all in-person and virtual visits
* No changes in medication or major surgical procedures anticipated for the trial
* Able to identify someone to accompany from the research unit at the end of drug administration day or agreement to have a study team member accompany them from the research unit

Exclusion Criteria:

* A health condition that makes this study unsafe or unfeasible, determined by study physicians
* Use of medication, vitamins, or supplements and unwilling or unable to discontinue medications that have problematic interactions with psilocybin
* Adulthood epilepsy or other seizure disorder
* Require supplemental oxygen
* Medical finding or diagnosis that would make participation in this trial unsafe

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in neural functional connectivity | Drug administration to 90 days following
  Measured by high-gamma coherence, cross-correlations, and Granger Causality

SECONDARY OUTCOMES:
Subjective changes in pain | Drug administration to 90 days following
  Measured by subjective pain scales

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, MD/PhD, Principal Investigator — University of California, San Francisco; Prasad Shirvalkar, MD/PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No